CLINICAL TRIAL: NCT06345157
Title: An ITAlian Observational, Multicenter, 12-month, Single-arm Study to Evaluate the Effectiveness and Safety of Treatment With Ofatumumab (Kesimpta®) in a pOpulation of RRMS Patients in a Real-world Setting - the ITAKOS Study
Brief Title: ITAKOS - Italian Observation, Multicenter, Prospective Study of Ofatumumab in RRMS Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157GIT02
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis,; Relapsing-Remitting,; RRMS,; ofatumumab
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — ofatumumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sample of whole blood to evaluate KREC, TREC and B and T cells subset. Sample of Serum to evaluate NfL.

GROUPS / COHORTS (1):
- Ofatumumab: Patients treated with Ofatumumab
  Interventions: Drug: Ofatumumab

INTERVENTIONS:
Drug: Ofatumumab — This is an observational study. There is no treatment allocation. The decision to initiate treatment with ofatumumab (Kesimpta®) will be based solely on clinical judgement and according to the SmPC and AIFA reimbursement criteria.
  Other Names: Kesimpta

SUMMARY:
Study to evaluate the effectiveness of ofatumumab in Italian RRMS patients in the real-life setting.

DETAILED DESCRIPTION:
Prospective real-world data on ofatumumab is still very limited. For this reason, the main aim of this study is to investigate the impact of ofatumumab in a population of Italian RRMS patients in routine clinical practice to evaluate if ofatumumab is able in these conditions to provide relevant clinical benefits that comprehensively encompass anti-inflammatory activity (relapses), disability accumulation, cognitive impairment, fatigue symptoms and quality of life.

This is an observational, multicenter, single-arm, prospective study. Prospective data will be collected on patients newly treated with ofatumumab over an observational period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients ≥18 years old.
2. Patients diagnosed with RRMS (McDonald criteria 2017).
3. Patients newly treated with ofatumumab, for whom the decision to start treatment with the drug has already been taken independently from study inclusion, based on clinical practice and according to the SmPC and to AIFA reimbursement criteria and who already successfully qualified for treatment with ofatumumab (i.e., passed the screening procedure mandated by the SmPC and the Risk Management Plan (RMP) for this treatment).
4. Patient or a legal representative of the patient must provide written informed consent before any study assessment is performed.

Exclusion Criteria:

1. Patients outside the approved label of ofatumumab.
2. Pregnant and lactating women.
3. Patients with any clinical condition that may interfere with the subject's ability to cooperate and comply with the study procedures based on investigator's judgement.
4. Patients cannot participate in this non-interventional study if they also participate in an interventional trial.
5. Treatment with ofatumumab prior to inclusion in this study or after 7 days from baseline visit.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 RRMS patients newly treated with ofatumumab.
Sampling Method: Probability Sample
Enrollment: 378 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Annualized relapse rate (ARR) | 1 year
  Annualized relapse rate (ARR) after a maximum observation period of 12 months of ofatumumab treatment.
  ARR is the number of confirmed relapses in a year, calculated as the total number of relapses for all participants in the treatment group divided by the total participant-years of time in study.

SECONDARY OUTCOMES:
Proportion of patients with an improvement in SDMT (Symbol Digit Modality Test) | Baseline, month 6, month 12
  To evaluate absolute and relative frequencies of patients with an improvement in SDMT (Symbol Digit Modality Test). An improvement is defined as an increase in the score of 4 or more points from baseline.
  The SDMT measures the time to pair abstract symbols with specific numbers. The test requires elements of attention, visuoperceptual processing, working memory, and psychomotor speed. The score is the number of correctly coded items from 0-110 in 90 seconds. The total score provides a measure of the speed and accuracy of symbol-digit substitution. Higher scores indicate better performance.
Fatigue Severity Scale [FSS] | Baseline, month 3, month 6 and month 12
  Proportion of patients passing from "fatigued" (F) to "not fatigued" (NF), according to the Fatigue Severity Scale [FSS].
  FSS is a 9-statement interview with a 7-point scale response per statement, with higher scores indicating more fatigue. Patients with a mean FSS score ≥ 4 are considered fatigued (F), while those with a mean FSS score < 4 not fatigued (NF).
Quality of life parameters assessed by EQ-5D-3L | Baseline, 12 months
  EQ-5D-3L is a descriptive questionnaire comprising five dimensions regarding mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has three response levels of severity: no problems, some problems, extreme problems. The respondent is asked to indicate his/her health state by checking the box next to the most appropriate response level of each of the five dimensions.
Treatment satisfaction assessed by TSQM-9 | Month 6, month 12
  Treatment Satisfaction Questionnaire for Multiple Sclerosis (TSQM-9). The TSQM-9 is a validated tool, widely used, to measure treatment satisfaction that will be applied in the context of this study regarding Ofatumumab. The TSQM-9 uses nine of the 14 TSQM Version 1.4 items, not including five questions related to side effects of medication, and comprises three scales: the effectiveness scale, the convenience scale and the global scale. The TSQM-9 domain scores range from 0 to 100 with higher scores representing higher satisfaction on that domain.
Expanded Disability Status Scale (EDSS) | Baseline, month 12 months
  Proportion of patients with an improved, stable or worsened EDSS. For patients with a baseline EDSS of 0 to 1.5, no disability improvement was possible based on the protocol definition of an improvement; for patients with a baseline EDSS of ≥2 to 6 or ≥6.5 to 9.5, the criterion for disability improvement was a decrease in EDSS of ≤1 or ≤0.5, respectively For patients with a baseline EDSS of 0, the criterion for disability worsening was an increase in EDSS of ≥1.5, for patients with a baseline EDSS of 1 to 5 or ≥5.5, the criterion for disability worsening was an increase in EDSS of ≥1 or ≥0.5, respectively.
Variation of NfL in plasma | Baseline, month 6 and month 12
  Variation of Neurofilaments (NfL) in plasma of the patients
Adverse Events (AEs) | 12 months
  Exposure-adjusted proportion of patients with adverse events (AE) or serious adverse events (SAE) per 100 subject-years.
Discontinuation rates due to AE and/or other reasons | 12 months
  Discontinuation rates due to AE and/or other reasons

CONTACTS AND LOCATIONS:
Locations (29):
- Italy (29):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, L’Aquila, AQ
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Chieti, CH
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Catanzaro, CZ
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Foggia, FG
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Pozzilli, IS
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Ravenna, RA
  - Novartis Investigative Site, Reggio Calabria, RC
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Sassari, SS
  - Novartis Investigative Site, Trento, TN
  - Novartis Investigative Site, Orbassano, TO
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Treviso, TV
  - Novartis Investigative Site, Udine, UD
  - Novartis Investigative Site, Gallarate, VA
  - Novartis Investigative Site, Vicenza, VI
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Novara